CLINICAL TRIAL: NCT06213961
Title: The Effect of Pecka Kucha Presentation on Basic Life Support Training on the Knowledge and Practice Levels of Students Studying in Healthcare: Randomized Controlled Study
Brief Title: The Effect of Pecha Kucha Presentation for Basic Life Support Training on Students' Knowledge and Practices Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MAİDE YEŞİLYURT (Other)
Collaborators: Aksaray University (Other)
Responsible Party: Sponsor-Investigator, MAİDE YEŞİLYURT, lecturer doctor, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Myesilyurt3
Record Dates: First submitted 2023-12-27; First posted 2024-01-19 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Basic Life Support
Keywords: pecha kucha; basic life support; health science; student

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm trained with pecha kucha (Experimental): Before basic life support training is given to students, an introductory characteristics form and basic life support skill questions will be applied (pre-test). Skill questions will be administered immediately after the PK training presentation, which includes basic life support skills, is given to the students (Posttest 1), and 4 weeks later.
  Interventions: Other: pecha kucha education
- control arm (No Intervention): Before basic life support training is given to students, an introductory characteristics form and basic life support skill questions will be applied (pre-test). Immediately after the traditional powerpoint training presentation, which includes basic life support skills, is given to the students (Posttest 1), the skill questions will be administered again 4 weeks later.

INTERVENTIONS:
Other: pecha kucha education — Basic life support training to be given to students will be given by the pecha kucha presentation method.
  Arms: arm trained with pecha kucha

SUMMARY:
Basic Life Support (BLS) is the practice performed to ensure oxygenation of the lungs and pumping of blood from the heart without medication or medical intervention in a person whose breathing and/or heart has stopped (Tiryaki and Doğu, 2018). In the vast majority of out-of-hospital cardiac arrest cases, the chance of survival is very low. Therefore, early, accurate and effective first aid application is vital (Shahrakivahed et al. 2015). The low survival rates after cardiac arrest indicate that basic life support skills still need to be developed and proficiency maintained during cardiopulmonary resuscitation (CPR) (Everett-Thomas et al. 2016).

DETAILED DESCRIPTION:
Nowadays, with technological developments, the use of new presentation techniques in addition to the methods used to develop knowledge, skills and practices in health sciences education is becoming increasingly widespread .Pecha kucha (PK) is an innovative form of presentation used around the world. PK, derived from the Japanese word meaning "chat", helps present creative works with visual images. Pecha kucha is a compact and effective presentation method consisting of 20 slides, each presented in 20 seconds This "20×20" format, which requires careful editing and develops the use of critical communication skills, serves as an innovative and valuable tool that allows the presenter to dynamically and systematically present important information worth sharing to the audience. Thanks to Pecha Kucha, the presenter conveys the topic quickly and clearly without deviating from the essence of the topic. PK may be superior to traditional PowerPoint presentations in terms of learning function. PK is as effective as traditional PowerPoint presentations in retaining information. It is stated that with the pecha kucha method, information can be presented in a more concise way, without any difference in quality, compared to a longer PowerPoint presentation. PK presentation, including visual and narrative presentation, does not take more than 7-8 minutes. It is stated that teachers and students prefer this technique due to its good presentation quality, increased eye contact and visual appeal, and attractiveness. In the literature, there is a lack of studies examining the knowledge and application skills of students regarding BLS education given using the Pecha Kucha method. In addition to contributing to the existing literature, this research will also contribute to determining the effect of basic life support training given with Pecha Kucha, a current presentation technique, on the learning and practice level of students studying in the field of health services.

ELIGIBILITY:
Inclusion Criteria:

* Having a stoma for the first time,
* Able to speak and understand Turkish,

Exclusion Criteria:

* Having previously had a stoma,
* Having difficulty speaking and understanding Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-04-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Basic life support knowledge level of students | up to 4 weeks
  In the form that questions the knowledge and application levels of basic life support application, each correct answer/application given by the student will be evaluated as 1 point and the average score will be calculated. Students will be able to get a minimum of 0, a maximum of 10 points from the knowledge test, and a minimum of 0 and maximum 17 points from the checklist. Three expert opinions were taken to evaluate the suitability of the prepared forms.
Basic life support application level of students | up to 4 weeks
  In the form that questions the knowledge and application levels of basic life support application, each correct answer/application given by the student will be evaluated as 1 point and the average score will be calculated. Students will be able to get a minimum of 0, a maximum of 10 points from the knowledge test, and a minimum of 0 and maximum 17 points from the checklist. Three expert opinions were taken to evaluate the suitability of the prepared forms.

CONTACTS AND LOCATIONS:
Overall Officials: MAİDE YEŞİLYURT, Principal Investigator — Aksaray University
Locations (1):
- Aksaray University, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol
Time Frame: pretest-posttest-4 weeks after
Access Criteria: after the application is completed